CLINICAL TRIAL: NCT03165760
Title: Protective Mechanical Ventilation and Risk of Postoperative Complications in Abdominal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mongi Slim Hospital (Other)
Responsible Party: Principal Investigator, Mhamed Sami Mebazaa, professor head of the anesthesiology-ICU departement, Mongi Slim Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Mongi Slim OR
Record Dates: First submitted 2017-05-19; First posted 2017-05-24 (Actual); Last update posted 2017-05-24 (Actual); Status verified 2017-05

CONDITIONS: Ventilator-Induced Lung Injury; Mechanical Ventilation Complication; Postoperative Complications
Keywords: protective mechanical ventilation
MeSH Terms: conditions — Ventilator-Induced Lung Injury; Postoperative Complications

STUDY DESIGN:
Intervention Model Description: randomization is decided when patients are schedueld and according a randomization table
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): Vt = 8 ml/kg of PBW and PEEP = 4 cm H2O
- protective ventilation group (Experimental): Vt = 6ml/kg of PBW, PEEP = 10 and RM if disconnected
  Interventions: Procedure: protective ventilation

INTERVENTIONS:
Procedure: protective ventilation — the aim of the intervention is to ovoid Ventilator induced lung injury and inflammatory stress
  Arms: protective ventilation group

SUMMARY:
Randomized controlled trial, comparing two groups of 40 patients each scheduled for open major abdominal surgery. The intervention group was ventilated with a protective strategy consisting on a low Tidal volume (Vt) (6ml/kg of predicted body weight (PBW)), positive end expiratory pressure (PEEP) = 10 cm H2O and recruitment manoeuvres (RM) after disconnection from the ventilator, the control group had classic ventilation (Vt = 8 ml/kg of PBW, PEEP = 4 cmH2O and no RM).

DETAILED DESCRIPTION:
This randomized controlled trial, was approved by the institutional ethics committee of our hospital. Informed consent was obtained from all the participants before randomization. Investigators included 80 patients (40 in each group), ASA I or II, planned for open abdominal surgery lasting more than 2 hours under general anesthesia.

Patients were not included if they had specially acute respiratory disease, severe asthma or emphysema, sleep apnea syndrome, septic shock and body mass index (BMI) < 16 or > 35 Kg/m2. Participants were excluded in case of serious peroperative anesthetic complications or hemorrhagic shock.

Primary endpoint was postoperative pulmonary complications occurring within the first 7 days after surgery (defined as hypoxemia, Broncho-pneumopathy, pulmonary infiltrate, acute respiratory distress syndrome, atelectasis, pleural effusion).

Secondary endpoints for all participants were intra-operative complications (change in SpO2 when dropped less than 90%, hypotension <90 mmHg lasting more than 3 min, need for vasopressor administration, new arrhythmia), postoperative extrapulmonary complications (septic shock, postoperative surgical complications, heart disease complications). Investigators recorded for all participants length of hospital stay and mortality rate were .

Investigators randomly allocated patients before entering to the operating room to:

* Control Group (CG): patients ventilated with Vt of 8 ml/kg of predicted body weight (PBW), a low level of PEEP (4 cm H2O) without RM.
* Protective Ventilation Group (PVG): patients ventilated with a low Vt of 6 ml/Kg of PBW, a high level of PEEP (10 cm H2O), RMs applied after intubation, before extubation and in case of disconnection from the ventilator.

Other ventilation settings, type of anesthesia, fluid administration and post operative pain management were standardized.

In the postoperative period, investigators daily assessed clinical examination and arterial blood gas if pulse oximetry dropped. For all participants, a chest X ray, blood count creatinine and C reactive protein were done at day 1 and day 3.

Data were presented as means and standard deviation [SD] or frequencies. Statistical analyses were performed using SPSS statistical software version 20.0. A p-value of 0.05 was considered significant.

ELIGIBILITY:
Inclusion Criteria:

* ASA I or II, planned for open abdominal surgery lasting more than 2 hours under general anesthesia

Exclusion Criteria:

* Patients were not included if they had specially acute respiratory disease, severe asthma or emphysema, sleep apnea syndrome, septic shock and BMI < 16 or > 35 Kg/m2. They were excluded in case of serious peroperative anesthetic complications or hemorrhagic shock.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Postoperative pulmonary complications | Postoperative pulmonary complications within the first 7 days after surgery
  Postoperative pulmonary complications occurring within the first 7 days after surgery (defined as hypoxemia, Broncho pneumopathy, pulmonary infiltrate, acute respiratory distress syndrome, atelectasis, pleural effusion)

IPD SHARING:
Plan to Share IPD: No